CLINICAL TRIAL: NCT00182234
Title: A Study of the Effectiveness of Specialist Oncology Nursing Case Management in Improving Continuity of Supportive Cancer Care in the Community (SONICS)
Brief Title: SONICS - Effectiveness of Specialist Oncology Nursing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Ministry of Health and Long Term Care (Other Government)
Responsible Party: Dr. Jonathan Sussman, Hamilton Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 74867; CIHR - 74867; MOHLTC - 04171
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Continuity of Care; Quality of Life
Keywords: unmet supportive care needs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Community Interlink Program — The study intervention is a referral to a specialized oncology nursing program. The standardized care provided by this program includes comprehensive assessment and care planning specific to breast and colorectal cancers during the initial phases of treatment, with a minimum of two home visits. Through consultation with the patient, nurses either provide direct (non-medical) care to address needs identified and/or coordinate linkage to services in the community.
  Other Names: Interlink Community Cancer Nurses

SUMMARY:
This research project will address the issue of gaps in continuity of supportive care for cancer patients during the early phases of the disease trajectory that result in unmet needs and unnecessary morbidity. The investigators intend to study the impact of a specialized cancer-nursing program, Interlink Community Cancer Nurses (Interlink) on patient outcomes. Impact will be assessed directly using a validated measure of continuity of care from the patients' perspective and validated measures of key supportive care patient outcomes including unmet needs, distress, uncertainty in illness, and quality of life, in a randomized trial.

DETAILED DESCRIPTION:
Main Research Question: Does community-based specialist oncology nursing case management improve continuity of cancer care and lead to fewer unmet cancer patient needs?

Why this research is important: This research proposal addresses the issue of gaps in continuity of supportive care for cancer patients during the early phases of the disease trajectory that result in unmet needs and unnecessary morbidity, prior to entry into a formalized cancer care system (e.g., a regional cancer centre or hospital with a cancer treatment program). This initial diagnostic period of cancer is associated with significant stress, anxiety and uncertainty that can impact upon overall quality of life for all types of cancer. These problems are further exacerbated by waiting times of up to 16 weeks between diagnosis and attendance in a formalized cancer treatment system. During this time patients will face a fragmented supportive care service system resulting in a substantial number of patients reporting unmet needs and distress. These care gaps have significant implications considering that 38% of women and 41% of men will develop cancer during their lifetime and that cancer incidence continues to rise with an estimated 139,000 new cases in Canada (over 54,000 of these in Ontario) in 2003. There has been growing interest in nursing models to address these gaps in supportive cancer care but at this time there is not sufficient high quality evidence upon which to base policy decisions to support the widespread introduction of this type of model. The results of this study will be very important for policy development for community cancer care in Ontario and in other provinces in Canada.

What is being studied: We will study the impact of a specialized nursing intervention (Interlink) on patient outcomes early in the disease trajectory. Impact will be assessed directly using validated measures in a randomized controlled trial design. These measures will include: continuity of care, unmet needs, psychological distress, uncertainty in illness, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed breast or colorectal cancer.
* In the initial stages of surgical consultation within the randomized surgical practices.
* Not had previous or concomitant malignancies (except for: non-melanoma skin cancer, or carcinoma in situ of the cervix).
* Have been informed of cancer diagnosis by the surgical office.
* Reside in the Interlink adult program service area.
* Legally able to provide informed consent (18 years of age or older).
* Able to speak and read English.
* Patients from an intervention designated practice, must agree to referral to Interlink and to receiving an in-home needs assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2005-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Difference in unmet supportive care needs between intervention and control group | 2 to 3 weeks after baseline; 8 to 10 weeks after baseline
Difference in continuity of care between intervention and control group | 2 to 3 weeks after baseline; 8 to 10 weeks after baseline
Difference in quality of life between intervention and control group | 2 to 3 weeks after baseline; 8 to 10 weeks after baseline

SECONDARY OUTCOMES:
Difference in uncertainty in illness between intervention and control group | 2 to 3 weeks after baseline; 8 to 10 weeks after baseline
Difference in use of resources between intervention and control group | 2 to 3 weeks after baseline; 8 to 10 weeks after baseline
Acute stress following surgery | 8 to 10 weeks after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Sussman, MD, CCFP, FRCP (c), MSc, Principal Investigator — Supportive Cancer Care Research Unit

REFERENCES:
- [Derived] Sussman J, Bainbridge D, Whelan TJ, Brazil K, Parpia S, Wiernikowski J, Schiff S, Rodin G, Sergeant M, Howell D. Evaluation of a specialized oncology nursing supportive care intervention in newly diagnosed breast and colorectal cancer patients following surgery: a cluster randomized trial. Support Care Cancer. 2018 May;26(5):1533-1541. doi: 10.1007/s00520-017-3981-4. Epub 2017 Nov 30. PMID 29189967